CLINICAL TRIAL: NCT06152224
Title: Comparison of the Duration of Use of the Leva® Pelvic Health System in Women With Fecal Incontinence
Brief Title: Use of the LEVA® Pelvic Health System for Fecal Incontinence
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-1304; A532810 (Other: UW- Madison); Protocol Version 10/1/2024 (Other: UW - Madison); SMPH/OBGYN BENIGN GYN (Other: UW - Madison)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Fecal Incontinence
Keywords: anal incontinence; accidental bowel leakage; pelvic health system
MeSH Terms: conditions — Fecal Incontinence; Encopresis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 8 week use of Leva (Experimental)
  Interventions: Device: The Leva Pelvic Health System
- 16 week use of Leva (Active Comparator)
  Interventions: Device: The Leva Pelvic Health System

INTERVENTIONS:
Device: The Leva Pelvic Health System — The Leva Pelvic Health System includes an intra-vaginal device that pairs with a smartphone application to provide real-time visual feedback about pelvic floor muscle performance during usage.

SUMMARY:
The goal of this clinical trial is to learn about how the duration of use of The Leva Pelvic Health System® affects treatment of fecal incontinence in women. The main question it aims to answer is to test whether use of the The Leva Pelvic Health System® for 8 weeks is as good as using it for 16 weeks.

Participants will complete surveys, and use the Leva device.

DETAILED DESCRIPTION:
This study will assess whether 8 weeks of use of the Leva Pelvic Health System (Leva) is non-inferior to 16 weeks of use for the treatment of chronic fecal incontinence (symptoms >/= 3 months) in adults with a vagina. Participants will be instructed to complete pelvic floor muscle training using the Leva for 8 or 16 weeks.

The hypothesis is that 8 weeks of use of Leva is non-inferior to 16 weeks of use, assessed by a validated FI symptom severity survey. Surveys will be completed at 0 weeks, 16 weeks, and 24 weeks. Long-term surveys will be completed at 1 year and 2 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥ 18years, assigned female at birth
* Fecal incontinence, defined as any uncontrolled loss of liquid or solid fecal material that occurs at least monthly over the last 3 months that is bothersome enough to desire treatment
* Able to stand to perform daily training for at least 3 minutes
* Able to speak and read English due to Leva smartphone application availability in only English at this time
* Have an email address, owns a smartphone, and can download an app

Exclusion Criteria:

* Inability to tolerate insertion of vaginal device (e.g., vaginal agenesis, vaginal stenosis, unremitting pelvic pain, within 12 weeks postpartum)
* Current diagnosis of colorectal or anal malignancy
* Diagnosis of uncontrolled inflammatory bowel disease
* Current rectovaginal fistula or cloacal defect
* Rectal prolapse (mucosal or full thickness)
* Inability to utilize smart phone technology ("app" use)
* Chronic Stool Types 6 or 7
* Fecal impaction by exam
* Stage 4 pelvic organ prolapse
* Concurrent supervised anal sphincter exercise/pelvic floor muscle training with or without biofeedback
* Presence of sacral neuromodulator
* Pelvic floor surgery (including anal sphincteroplasty) within the past 3 months
* Currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dobie Giles, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Started | 19 | 19
8 Week Follow-up | 18 | 18
16 Week Follow-up Surveys | 18 | 18
16 Week Follow-up Visit | 18 | 17
Completed 24 Week Time Point | 18 | 18
Completed | 0 | 0
Not Completed | 19 | 19
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — On Follow Up | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (13.7) | 60.4 (17.0) | 62.9 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Brinks Score [Median (Inter-Quartile Range); unit: units on a scale] — Brink Scale measures pelvic floor muscle strength, scored from 1-4 in 3 areas:
  * Pressure where 1 is no response and 4 is a strong squeeze
  * Vertical Displacement where 1 is none and 4 is whole fingers pulled in
  * Duration Contraction where 1 is no contraction and 4 is greater than 3 seconds
  units on a scale
    Pressure | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 2.0]
    Vertical Displacement | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
    Contraction Duration | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (7.9) | 31.5 (9.4) | 29.3 (8.8)
Pelvic Organ Prolapse (POP-Q) [Count of Participants; unit: Participants] — * Stage 1: Most distal prolapse is more than 1 cm above the hymen
  * Stage 2: Most distal prolapse is between 1 cm above and 1 cm below the hymen
  Participants
    Stage 1 | 9 | 10 | 19
    Stage 2 | 10 | 9 | 19
Vaisey Score [Mean (Standard Deviation); unit: units on a scale] — A measure of incontinence scored from 0 (perfect continence) to 24 (totally incontinent)
  units on a scale | 13.3 (4.3) | 12.5 (4.3) | 12.9 (4.3)
Bristol Stool Scale [Count of Participants; unit: Participants] — Description of stool between 1-7
  * Type 1: separate hard lumps, like nuts (hard to pass)
  * Type 2: sausage shaped but lumpy
  * Type 3: like a sausage but with cracks on the surface
  * Type 4: like a sausage or a snake, smooth and soft
  * Type 5: soft blobs with clear edges, (passed easily)
  * Type 6: fluffy pieces with ragged edges, a mushy stool
  * Type 7: watery, no solid pieces, entirely liquid
  Participants
    Type 1 | 0 | 3 | 3
    Type 2 | 1 | 1 | 2
    Type 3 | 0 | 3 | 3
    Type 4 | 11 | 4 | 15
    Type 5 | 4 | 3 | 7
    Type 6 | 3 | 5 | 8
    Type 7 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Vaizey Score to Compare Effectiveness of Improving Fecal Incontinence Between 8 Weeks and 16 Weeks of Use
Description: Treatment response as length of use on symptom improvement at 16 weeks (comparing 8 weeks vs 16 weeks of use of Leva) as assessed by Vaizey Score, score ranges from 0-24, higher scores indicate more severe symptoms. A difference of -4.3 ± 3 is expected at 8 weeks and 16 weeks (compared to baseline), with an allowable difference of 1.
Time Frame: Baseline to 16 weeks
Population: one participant withdrew, one participant was lost to follow up at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Number analyzed (Participants) | 19 | 19
score on a scale
  baseline | 13.3 (4.3) | 12.5 (4.3)
  16 weeks: number analyzed (Participants) | 18 | 18
  16 weeks | 9.0 (5.4) | 7.5 (4.4)
Statistical Analysis 1: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; change from baseline; Test type: Equivalence — Power analysis was determined based on a 4.3 point improvement on the Vaizey score in both groups. With an allowable difference of 1 point between randomized groups, standard deviation = 3, margin = 4.3, power = 0.8, alpha = 0.05, attrition = 25 percent; p = 0.918, t-test, 2 sided — a priori threshold 0.05; continuous outcome; Mean Difference (Final Values) = -4.3, Standard Deviation 3

2. Secondary Outcome: Change in Fecal Incontinence Severity
Description: Using St. Mark's Incontinence score, score ranges from 0-24, higher scores indicate more severe symptoms.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Cumulative Adherence Correlation With Change in St. Mark's Score
Description: Adherence as a percentage of all expected exercise sessions correlated with change in St Mark's Incontinence Score (1-24)
Time Frame: Baseline to 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Patient Satisfaction and Usability of the Smartphone Application Component of the Leva Pelvic Health System
Description: Measured through the mHealth App Usability Questionnaire. In this questionnaire, 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree. To determine the usability of an app, calculate the total and determine the average of the responses to all statements. The higher the overall average, the higher the usability of the app.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Change in Fecal Incontinence From Baseline to 24 Weeks After 8 or 16 Weeks of Treatment
Description: Treatment response as length of use on symptom improvement at 24 weeks (comparing 8 weeks vs 16 weeks of use of Leva) as assessed by St Mark's (Vaizey) scores.
Time Frame: Baseline to 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Change in Pelvic Organ Prolapse Quantification System (POP-Q)
Description: The POP-Q system is an objective, site-specific system used to describe, quantify, and stage pelvic support. Measurements are rated as Stage 0-Stage 4, with Stage 4 being complete prolapse.
Time Frame: Baseline to 16 weeks
Population: one participant withdrew, one participant was lost to follow up at 16 weeks, one participant completed 16-week surveys but did not follow up for in person visit
Measure: Count of Participants; unit: Participants
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Number analyzed (Participants) | 19 | 19
Participants
  Baseline: Stage 1 | 9 | 10
  Baseline: Stage 2 | 10 | 9
  Baseline: Stage 3 | 0 | 0
  16 weeks: number analyzed (Participants) | 18 | 17
  16 weeks: Stage 1 | 9 | 10
  16 weeks: Stage 2 | 8 | 7
  16 weeks: Stage 3 | 1 | 0
Statistical Analysis 1: Comparison: 8 Week Use of Leva; change from baseline; Test type: Equivalence — Power analysis was determined based on a 3 point improvement on the Vaizey score in both groups. With an allowable difference of 1 point between randomized groups, type I error level = 0.05, power = 0.8, and standard deviation of outcome of 4; p = 0.801, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 2: Comparison: 16 Week Use of Leva; change from baseline; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.317, t-test, 2 sided — a priori threshold 0.05; continuous outcome

7. Secondary Outcome: Change in Brink Scale Score: Pressure
Description: The Brink scale evaluates 3 PFM contraction variables: vaginal pressure or muscle force, elevation or vertical displacement of the examiner's fingers, and duration of contraction. Each muscle contraction variable is rated on a 4-point ordinal scale (1-4). Higher scores indicating greater strength.
Time Frame: Baseline to 16 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Number analyzed (Participants) | 19 | 19
score on a scale
  Baseline | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 3.0]
  16 weeks: number analyzed (Participants) | 18 | 17
  16 weeks | 3.0 [3.0 to 3.0] | 4.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: 8 Week Use of Leva; change from baseline Brink Score: Pressure; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 2: Comparison: 16 Week Use of Leva; change from baseline in Brink Score: Pressure; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome

8. Secondary Outcome: Change in Brink Scale Score: Vertical Displacement
Description: as for outcome 7
Time Frame: Baseline to 16 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Number analyzed (Participants) | 19 | 19
score on a scale
  Baseline | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  16 weeks: number analyzed (Participants) | 18 | 17
  16 weeks | 2.5 [2.0 to 4.0] | 4.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: 8 Week Use of Leva; Change from baseline in Brink Score: Vertical Displacement; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 2: Comparison: 16 Week Use of Leva; change from baseline in Brink Score: Vertical Displacement; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome

9. Secondary Outcome: Change in Brink Scale Score: Duration Contraction
Description: as for outcome 7
Time Frame: Baseline to 16 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
Number analyzed (Participants) | 19 | 19
score on a scale
  Baseline | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  16 weeks: number analyzed (Participants) | 18 | 17
  16 weeks | 4.0 [3.0 to 4.0] | 4.0 [4.0 to 4.0]
Statistical Analysis 1: Comparison: 8 Week Use of Leva; change from baseline in Brink Score: Duration Contraction; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 2: Comparison: 16 Week Use of Leva; change from baseline in Brink Score: Duration Contraction; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, t-test, 2 sided — a prior threshold 0.05; continuous outcome

10. Secondary Outcome: Change in Stool Consistency
Description: Use the Bristol Stool Scale to evaluate stool consistency. Ranges from Type 1 to Type 7, where Type 1 is hardest consistency and Type 7 is entirely liquid.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

11. Secondary Outcome: Change in Fecal Incontinence Quality of Life (FIQoL)
Description: Use FIQoL scale, in which participants rate questions about how often an issue is a concern, and how much they agree with statements on a scale of 1-5. Higher scores indicate lower quality of life.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

12. Secondary Outcome: Change in Sexual Function (PISQ-IR)
Description: PISQ-IR is a 20 item survey, where higher scores indicate lower sexual function.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

13. Secondary Outcome: Patient Global Impression of Improvement (PGI-I)
Description: PGI-I is a 2 question qualitative survey in which participants state their satisfaction and perception of improvement.
Time Frame: 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

14. Secondary Outcome: Patient Satisfaction (PGI-I)
Description: PGI-I is a 2 question qualitative survey in which participants state their satisfaction and perception of improvement.
Time Frame: 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

15. Secondary Outcome: Estimated Percentage of Change
Description: Qualitative question in which participants state their estimate of how much better they are, on a scale from 0% (no better) to 100% (completely better).
Time Frame: 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

16. Secondary Outcome: Change in Global Pelvic Floor Symptoms
Description: Use the Pelvic Floor Distress Inventory (PFDI-20) to evaluate change in pelvic floor symptoms. It is a 20 item survey with a range from 0-100 where higher scores indicate greater symptoms.
Time Frame: Baseline to 16 and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

17. Secondary Outcome: Evaluate Self-continuation of Pelvic Floor Muscle Exercises
Description: Participant self-report on whether and how often they continued the pelvic floor muscle exercises.
Time Frame: Baseline and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

18. Secondary Outcome: Number of Cumulative Adverse Events
Description: Systematic assessment of all adverse events over the course of the study, reported as a number of total AEs.
Time Frame: Baseline and 24 weeks, long term follow up at 1 and 2 years
Reporting Status: Not Posted

19. Secondary Outcome: mHealth App Usability Questionnaire (MAUQ)
Description: MAUQ is an 18-item survey scored on a 7 point likert scale from 1 (disagree) to 7 (agree) with higher scores indicative of higher usability.
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- All Participants: Summary data for all participants together.
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva | All Participants
Number analyzed (Participants) | 18 | 18 | 36
score on a scale
  Q1. The app was easy to use | 6.0 [5.0 to 7.0] | 7.0 [6.0 to 7.0] | 7.0 [6.0 to 7.0]
  Q2. It was easy for me to learn to use the app | 7.0 [6.0 to 7.0] | 7.0 [7.0 to 7.0] | 7.0 [6.0 to 7.0]
  Q11. I would use this app again | 7.0 [4.0 to 7.0] | 7.0 [6.0 to 7.0] | 7.0 [5.5 to 7.0]
  Q12. Overall, I am satisfied with this app | 6.0 [6.0 to 7.0] | 7.0 [6.0 to 7.0] | 6.5 [6.0 to 7.0]
  Q15. The app helped me manage my health effectively | 6.0 [3.0 to 7.0] | 6.0 [5.0 to 7.0] | 6.0 [3.5 to 7.0]
Statistical Analysis 1: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; Q1. The app was easy to use; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.035, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 2: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; Q2. It was easy for me to learn to use the app; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.063, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 3: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; Q11. I would use this app again; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.587, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 4: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; Q12. Overall, I am satisfied with this app; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.107, t-test, 2 sided — a prior threshold 0.05; continuous outcome
Statistical Analysis 5: Comparison: 8 Week Use of Leva vs 16 Week Use of Leva; Q15. The app helped me manage my health effectively; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.486, t-test, 2 sided — a prior threshold 0.05; continuous outcome

ADVERSE EVENTS:
Time Frame: up to 16 weeks (for primary outcome at the time of reporting)
Arm/Group | 8 Week Use of Leva | 16 Week Use of Leva
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 8 Week Use of Leva (N=19) | 16 Week Use of Leva (N=19)
Sciatic Pain (Nervous system disorders) | 1 | 0
Pelvic Pain with Urination (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT06152224/Prot_SAP_000.pdf